CLINICAL TRIAL: NCT03995524
Title: Perceived Spasticity and Treatment Satisfaction Among Stroke Survivors Over the Course of a Complete Treatment Cycle With Botulinum Neurotoxin A (BoNT-A): an Ethnographic Study.
Brief Title: Spasticity and Treatment Satisfaction Among Stroke Survivors
Acronym: REBOT
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: F-FR-52120-258
Record Dates: First submitted 2019-05-29; First posted 2019-06-24 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Spasticity as Sequela of Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate, through ethnography, changes in symptom burden and disability and their effects/interference on patient functioning, ability to perform activities of daily living (ADL) and quality of life (QoL) throughout the duration of one BoNT-A treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of post-stroke spasticity more than three months prior to inclusion
* At least 6 months on treatment (or two treatment cycles) with BoNT-A injections for spasticity according to the decision of the physician
* Previous BoNT-A injection cycles did not last for more than 16 weeks
* Ambulatory (use of walking aids is acceptable)

Exclusion Criteria:

* Neurological disorder other than stroke
* Spasticity-specific treatment changes within 3 months prior to inclusion
* Patients who had undergone neurolysis or surgery to the affected limb within 6 months
* Concurrent participation in a clinical trial for the treatment of spasticity

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 40 Adults subjects (male or female) suffering from post-stroke spasticity (the US, UK, France, and Italy), who are treated with BoNT-A in the course of routine clinical practice for focal spasticity
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Degree of functional limitations in daily life activities | monthly for 12 Weeks, or until end of injection cycle whichever occurs first
  Degree of functional limitations in daily life activities (i.e. physical functioning) associated with post-stroke spasticity as assessed by using WHODAS parameters, and identification of their characteristics and changes over time
Health status in subjects with post-stroke spasticity | weekly for 12 Weeks, or until end of injection cycle whichever occurs first
  Health status in subjects with post-stroke spasticity as assessed by using EQ-5D-5L parameters, and identification of their characteristics and changes over time
Severity of Pain | 12 weeks
  Severity of Pain as per EQ-5D-5L and a sliding scale. This is a descriptive scale that covers 5 dimensions: mobility, self-care, usual activities,pain/discomfort and anxiety/depression. the scale consist of 5 levels, where level one corresponds to "no problems" and level 5 corresponds to "extreme problem".

SECONDARY OUTCOMES:
Burden of spasticity/treatment | Opening interview and ending qualitative interviews, ethnography data which will be provided at discretion of patient/caregiver for 12 weeks or duration of treatment, whichever occurs first, may also support these qualitative analyses
  Themes/domains related to the everyday life experiences of subjects with post-stroke spasticity (e.g. burden disease/treatment) through qualitative analysis of in-depth open-ended interviews
Patients' satisfaction | weekly for 12 weeks or until end of injection cycle whichever occurs first. Opening and closing interview will also explore this
  Subjects Report of Satisfaction with Treatment and their perception/desire of more tailored treatment options
Comparison of feedback between caregivers and stroke survivors | opening ( before week 1) and ending ( 2 weeks after end of injection cycle) qualitative interviews
  Agreement between the themes elicited from semi-structured interviews between caregivers and subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Paris, France